CLINICAL TRIAL: NCT03551405
Title: 4D Cone Beam CT Reconstruction for Radiotherapy Via Motion Vector Optimization
Status: Terminated | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 082014-030
Record Dates: First submitted 2018-05-18; First posted 2018-06-11 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensity accuracy: The difference of the HU values in corresponding ROIs in the two image sets will be compared with zero using one sample t-test.
  In addition, we will also use these patient cases to test the computational efficiency of our algorithm. Based on our preliminary study, it is expected that the computation time will be 5~10 sec per phase. The reconstruction time will be recorded in these patient cases and will be assessed.
  Interventions: Radiation: CBCT scan

INTERVENTIONS:
Radiation: CBCT scan — CBCT is a standard image guidance procedure for patient setup in image-guided radiation therapy at the Department of Radiation Oncology, UTSW. Our study will deliver three additional CBCT scans to each patient in only one fraction. These additional scans will increase radiation doses to the patients, which elevate the radiation-associated risks of secondary cancer.The other risk involved in this study is a possible violation of patient confidentiality. The imaging data will be completely anonymized, since the patient related information is not needed for this study.

SUMMARY:
To validate a new 4D Cone Beam CT (4DCBCT) reconstruction algorithm that was developed in our research group recently in terms of its geometry and intensity accuracy through real patient studies. Dose calculation found out in this study will not be used on the subject

DETAILED DESCRIPTION:
Before patient studies, we will have conducted experimental studies on a lung phantom.

The purpose of this step is to comprehensively evaluate the system performance and gain confidence prior to its applications to real patient cases. We will operate the phantom to simulate motion patterns with different motion amplitude/frequency. 4DCBCT images will be reconstructed using our method and the conventional FDK algorithm. The validation will focus on two aspects: HU value accuracy and anatomy location accuracy.

Imaging dose in these scans will be also measured in phantom studies to make sure the radiation dose level is acceptable for patient studies. adiation dose level is acceptable for patient studies.

After testing the reconstruction algorithm on phantoms, we will move on to real patient cases. We will conduct patient studies on lung cancer patients treated under Image Guided Radiation Therapy (IGRT) at Department of Radiation Oncology, UT Southwestern Medical Center. CBCT projection data will be collected (4 gantry rotations, each within 1 minute) in only one treatment fraction. 4DCBCT images will be reconstructed from the current standard FDK algorithm using all the projection data, and from our system using data only in the first gantry rotation. Patient 4DCT image will also be used, which have been acquired during treatment planning stage per standard treatment protocol at UTSW.

The image quality of our 4DCBCT will be assessed in two aspects:

1) geometry accuracy, by comparing selected anatomical landmark locations with those in 4DCBCT reconstructed by the FDK algorithm. 2) HU accuracy, by comparing HU values in selected regions of interest (ROIs) with those in 4DCT.

The 4DCT images will be extracted from radiation therapy information system MOSAIQ.

The CBCT projection data will be exported from a computer that controls the image acquisition system

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have been diagnosed with lung cancer, and are treated at Department of Radiation Oncology, UTSW.
2. Patients are greater than 18 years of age.
3. Patients understand a written informed consent document and are willing to sign the consent form.

Exclusion Criteria:

1. Women who are pregnant or trying to get pregnant
2. Children (under age of 18)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by physician co-investigator during CT-simulation stage. One of the investigators or research coordinators will verbally explain the study to the patient.
  It will be clearly explained that patient's treatment will not be modified based on the data collected in this study. If the patient agrees to participate, an informed consent form will be signed by both the patient and the investigator/research coordinator and a copy of the signed form will be given to the patient. All of the key investigators and research coordinators in this project are experienced in clinical studies and clinical trials and have undergone appropriate protection of human research subjects training and HIPAA training.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Potential Benefits: | 10 years
  There is no direct benefit from the study to the subjects. All participants will be clearly informed about this. The individual patient's treatment will not be changed based on the data collected from these procedures.The study will use the CTCAE version 4.0 for reporting of acute and late adverse events related to Lung will be reported by the physician through exam/assessment during research visit, encompassing events since last research visit. Upon completion, the project will lead to an accurate and safe 4DCBCT imaging procedure for patient positioning to facilitate lung IGRT treatment.where the image quality is much improved compared to current standard 4DCBCT method and the scan time and hence radiation dose is greatly reduced.

SECONDARY OUTCOMES:
Risk/Benefit Ratio: | 10 years
  The benefits greatly outweigh the risks in this study. Considering the patient typically receives 60~80 Gy radiation dose for radiation treatment, the additional radiation dose from three additional CBCT scans is very small, and the risk is minimal. We have also established a set of procedures to ensure the safe use of medical data to protect patient confidentiality.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Jia, PHd — UTSW Radiation Oncology
Locations (1):
- UT Southwestern Medical Centre, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided